CLINICAL TRIAL: NCT07021287
Title: Effect of Different Cold Therapy Programs on NRS(Numerical Rating Scale),ROM(Range of Motion),GCQ(General Comfort Questionnaire), and Swell in Patients Received Total Knee Arthroplasty Operation
Brief Title: Effect of Different Cold Therapy Programs in Patients Received Total Knee Arthroplasty Operation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY-2024-218
Record Dates: First submitted 2025-04-02; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Arthroplasty
Keywords: cold therapy;; NRS; GCQ; ROM;
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mixed ice and water, continuous ice application (Experimental): after returning to the ward, the ice pack was placed on the knee joint for 24 hours, and the ice pack was replaced every 3 to 4 hours, if it melted, replaced immediately.
  Interventions: Other: mixed ice and water, continuous ice application
- mixed ice and water, intermittent ice compress (Experimental): within 72 hours after operation, the ice compress time was 30 minutes each time, the interval time was 2 hours, 3 times a day
  Interventions: Other: mixed ice and water, intermittent ice compress
- full ice, continuous ice compress (Experimental): after returning to the ward, the ice pack was placed on the knee joint for 24 hours, and the ice pack was replaced every 3 to 4 hours, if it melted, replaced immediately
  Interventions: Other: full ice, continuous ice compress
- full ice, intermittent ice compress (Experimental): within 72 hours after operation, the patients were given ice compress for 20 minutes each time, with an interval of 2 hours, 3 times a day.
  Interventions: Other: full ice, intermittent ice compress

INTERVENTIONS:
Other: mixed ice and water, continuous ice application — the ice pack was placed on the knee joint immediately after returning to the ward for 24 hours, and the ice pack was replaced every 3 to 4 hours, if it melted, replaced immediately.
  Arms: mixed ice and water, continuous ice application
Other: mixed ice and water, intermittent ice compress — within 72 hours after operation, the patients were given ice compress for 20 minutes each time, with an interval of 2 hours, 3 times a day
  Arms: mixed ice and water, intermittent ice compress
Other: full ice, continuous ice compress — After returning to the ward, an ice pack should be placed on the knee for 24 hours. The ice pack should be replaced every 3-4 hours and replaced immediately if melted
  Arms: full ice, continuous ice compress
Other: full ice, intermittent ice compress — Within 72h after surgery, the patient applied ice for 20min each time, with an interval of 2h,3 times a day.
  Arms: full ice, intermittent ice compress

SUMMARY:
This study conducts clinical experiments on the form, temperature, frequency and other issues of cooling therapy, so as to provide scientific evidence for the practice of cooling therapy and improve the comfort and effect of cooling therapy, so as to achieve the goal of improving service and patient experience proposed by the National Health Commission.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a degenerative joint disease that severely impacts patients' quality of life, primarily manifesting as knee pain and restricted mobility [1]. According to the Osteoarthritis Diagnosis and Treatment Guidelines (2018 Edition) [1], the prevalence of symptomatic knee osteoarthritis in China is 8.1%. Total knee arthroplasty (TKA) is primarily indicated for elderly patients with severe late-stage KOA-related pain and functional impairment. TKA not only improves knee function and corrects deformities but also significantly enhances patients' quality of life. Research by Feng et al. [2] demonstrates a rapid increase in TKA cases in China, rising from 53,880 cases in 2011 to 374,833 cases in 2019-a 5.9-fold growth. However, moderate to severe postoperative pain following TKA remains a major challenge, adversely affecting rehabilitation, patient satisfaction, and clinical outcomes .

Current postoperative pain management strategies for TKA include pharmacological and non-pharmacological interventions. While pharmacological approaches are relatively well-established and effective, they carry side effects such as nausea, vomiting, dizziness, and dependency. Non-pharmacological interventions include cold therapy, localized elastic bandage compression, limb elevation, and early rehabilitation exercises [5-7]. Cold therapy, a simple and cost-effective physical intervention, involves applying ice packs or cold water to reduce skin temperature, thereby decreasing local tissue metabolism, promoting vasoconstriction, reducing edema and hematoma formation, and slowing nerve conduction to alleviate pain. Additionally, cold therapy mitigates local inflammatory responses and blood loss, effectively improving pain and patient comfort .

Existing studies on cold therapy at varying temperatures for TKA are limited, with significant discrepancies in recommended application durations . Excessively low temperatures risk superficial or deep tissue frostbite, nerve damage, and even deep vein thrombosis or necrosis, while insufficient cooling may compromise analgesic and anti-inflammatory efficacy . Although cold therapy is widely adopted post-TKA, critical parameters-such as modality, temperature, frequency, and duration-remain controversial in clinical practice.

This study aims to address these unresolved issues through a clinical trial, generating scientific evidence to optimize cold therapy protocols. The findings will enhance patient comfort and therapeutic outcomes, aligning with the National Health Commission's goals of improving healthcare services and patient experiences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years after primary total knee arthroplasty
* No history of open injury or prior surgery in the affected knee

Exclusion Criteria:

* Motor, sensory, or cognitive dysfunction
* History of mental disorders
* Coagulation abnormalities
* Chronic use of oral corticosteroids (>3 months)
* Cold hypersensitivity/allergy
* Withdrawal due to non-study-related reasons
* Thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale ，NRS | Day 1, Day2, Day 3
  ostoperative pain intensity will be evaluated using the Numerical Rating Scale (NRS) at 24 hours following total knee arthroplasty (TKA). The NRS is an 11-point scale ranging from 0 to 10, where 0 represents "no pain" and 10 indicates "the worst imaginable pain." Patients will self-report their pain level by selecting a numerical value corresponding to their perceived intensity. The scale is visually presented as a 10-cm horizontal line divided into 10 equal segments, with each segment labeled sequentially from 0 to 10.
general comfort questionnaire，GCQ | Day 1, Day2, Day 3
  GCQ was developed by the famous nursing scientist Kekaba. In 2004, it was sinicized by Chinese scholar Julixia et al. It is suitable for all kinds of people with discomfort. The scale contains four dimensions of physiology, psychology, environment and social culture, a total of 28 items, using 1-4 Likert scores, with 1 indicating "strongly disagree" and 4 indicating "strongly agree". The total scores range from 28 to 112. That is, patients were in low comfort (total score < 60), moderate comfort (60-90 points) and high comfort (> 90 points). Clinical research found that the scale had good reliability and validity (Cronbach's α coefficient was 0.893).
Joint range of motion (ROM), knee swelling | Day 1, Day2, Day 3
  Range of Motion (ROM)
  Range of Motion (ROM), also termed joint range of motion, refers to the maximum arc of movement achievable by a joint during motion. ROM is categorized into two types based on the force driving the movement:

CONTACTS AND LOCATIONS:
Overall Officials: Cheng li Yan, Bachelor, Principal Investigator — Study Principal investigatorThe Fourth Affiliated Hospital of Zhejiang UniversitySchool of Medicine
Locations (2):
- China (2):
  - 4th Affiliated Hospital, School of Medicine, ZhejiangUniversity, China, Yiwu, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No